CLINICAL TRIAL: NCT06255795
Title: The Efficacy and Safety of Chidamide, Anti-PD-1 Antibody in Combination With Pegaspargase Versus DDGP in the Treatment of Newly Diagnosed, Stage III to IV Extranodal Natural Killer/T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-NKTCL-3
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Extranodal Natural Killer T Cell Lymphoma
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; pegaspargase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chidamide, anti-PD1 antibody, and pegaspargase group (Experimental)
  Interventions: Drug: chidamide, anti-PD1 antibody, and pegaspargase
- DDGP (Active Comparator)
  Interventions: Drug: DDGP

INTERVENTIONS:
Drug: chidamide, anti-PD1 antibody, and pegaspargase — 6 cycles of pegaspargase 2500IU/m2 intramuscularly on day1, anti-PD1 antibody 200mg intravenously on day 2, chidamide 30mg biw orally, every 21 days.
  Arms: chidamide, anti-PD1 antibody, and pegaspargase group
Drug: DDGP — 6 cycles of pegaspargase 2500IU/m2 intramuscularly on day1, cisplatin 20mg/m2 intravenously on days 1 through 4, dexamethasone 15mg/m2 intravenously on days 1 through 5, gemcitabine 800mg/m2 on day 1 and day 8, every 21 days.
  Arms: DDGP

SUMMARY:
A multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of chidamide, anti-PD1 antibody, and pegaspargase versus dexamethasone, cisplatin, gemcitabine, and pegaspargase (DDGP) in the treatment of newly diagnosed, stage III to IV extranodal natural killer/T-cell lymphoma.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of chidamide, anti-PD1 antibody, and pegaspargase versus DDGP in the treatment of newly diagnosed, stage III to IV extranodal natural killer/T-cell lymphoma. Subjects will be randomly assigned 1:1 to chidamide, anti-PD1 antibody, and pegaspargase or DDGP regimen.

Patients in chidamide, anti-PD1 antibody, and pegaspargase group will receive 6 cycles of pegaspargase 2500IU/m2 intramuscularly on day1, anti-PD1 antibody 200mg intravenously on day 2, chidamide 30mg biw orally, every 21 days. Patients in DDGP group will receive 6 cycles of pegaspargase 2500IU/m2 intramuscularly on day1, cisplatin 20mg/m2 intravenously on days 1 through 4, dexamethasone 15mg/m2 intravenously on days 1 through 5, gemcitabine 800mg/m2 on day 1 and day 8, every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of NKTCL
* No previous anti-lymphoma treatment
* Age 14-70 years
* Ann Arbor stage III-IV
* At least one measurable/evaluable site after diagnostic biopsy before treatment start
* ECOG performance status of 0-2
* Adequate hematological and organ function; i.e. ANC >1000 cells /mmc, platelet counts > 50.000/mmc, Hemoglobin > 8 g/dl AST, ALT > 1.5 x ULN; serum bilirubin > 2x ULN (patient with Gilbert disease can be enrolled), Serum creatinine > 2 x ULN or creatinine clearance > 50ml/min
* Tumor tissue (fresh preferred, achievable tissue is also acceptable)
* For women of childbearing potential a negative pregnancy test on day 1 of cycle 1 and agree to adopt adequate measure to avoid pregnancy during study treatment and for at least one year from EOT.
* For men agreement to remain abstinent or to use barrier contraception
* Signed Informed consent

Exclusion Criteria:

* Confirmed histological diagnosis of aggressive NK cell leukemia
* Early stage disease (AA stage I-II)
* Evidence of suspect of CNS disease.
* Has an active autoimmune disease that has required systemic treatment in past 2-years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs), including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associate with antiphospholipid syndrome, wegener's granulomatosis, Sjogren syndrome, guillan barreè syndrome, multiple sclerosis, vasculitis or glomerulonephritis. The following exception are allowed: patients with autoimmune related hypothyroidism or type I diabetes mellitus who are on stable treatment. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Treatment with systemic immunosuppressive medications, including prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide and anti tumor necrosis factor (anti-TNF) agents within 2 weeks prior to cycle 1 day 1; inhaled corticosteroids are allowed.
* Active infection requiring systemic therapy
* History of (non-infectious) pneumonitis that required steroids; evidence of interstitial lung disease or active, non-infectious pneumonitis
* Significant cardiovascular disease, myocardial infarction in the previous 3 months, unstable arrhythmias, or unstable angina.
* History of other(s) infiltrating cancer(s) in the previous 3 years that were not treated with curative intent or who are still receiving anticancer therapy (including hormone therapy for breast or prostate cancer).
* HBsAg, HCV or HIV positivity. Positive serology is admitted for HBV and HCV but DNA/RNA test must be negative
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Pregnant or lactating women
* Administration of a live attenuated vaccine within 4 weeks before cyle 1 day 1. Patients must not receive live, attenuate vaccines, including influenza vaccines at any time during study.
* Other uncontrollable medical condition that may that may interfere the participation of the study

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival in the overall study population was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Percentage of Participants Achieving Meaningful Improvement in European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) | Baseline (pre-dose [Hour 0] on Cycle1 Day1), Cycle3 Day 1, end of treatment (up to Month 6), every 3 months 1st year, every 6 months 2nd year, and 12 months thereafter up to data cut-off, up to approximately 4 years (cycle length = 21 days)
  The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No